CLINICAL TRIAL: NCT01025817
Title: A 12 Month, Multi-center, Randomized, Open-label Non-inferiority Study Comparing Safety and Efficacy of Concentration-controlled Everolimus With Low Dose Tacrolimus to Mycophenolate Mofetil With Standard Dose Tacrolimus in de Novo Renal Transplant Recipients
Brief Title: Non-inferiority Study of Safety and Efficacy of Everolimus With Low Dose Tacrolimus to Mycophenolate Mofetil With Standard Dose Tacrolimus in Kidney Transplant Recipients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001AUS92
Record Dates: First submitted 2009-11-19; First posted 2009-12-04 (Estimated); Results first posted 2014-06-06 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-10

CONDITIONS: Kidney Transplant
Keywords: Kidney transplant; renal transplant; immunosuppression; mycophenolate mofetil; tacrolimus; everolimus
MeSH Terms: interventions — Everolimus; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Everolimus (EVR) & low dose of tacrolimus (Experimental): Everolimus (EVR) and tacrolimus treatment arm: Therapeutic drug monitoring of everolimus and tacrolimus was mandatory throughout the study. From Day 5 onwards, the everolimus 0.75 mg b.i.d. dose was increased if the trough level was < 3 ng/mL, or reduced if the trough level was > 8 ng/mL. Tacrolimus was initiated according to local practice. In this treatment arm, the tacrolimus dose was adjusted from Day 3 onwards, to a target whole blood trough concentration of 4 ng/mL to 7 ng/mL. From Month 2 until Month 6, the target tacrolimus trough level was 3 ng/mL to 6 ng/mL. After Month 6, the tacrolimus dose was adjusted in order to achieve a target trough level of 2 ng/mL to 5 ng/mL.
  Interventions: Drug: Everolimus and tacrolimus
- Mycophenolate mofetil & standard dose tacrolimus (Active Comparator): Mycophenolate mofetil and tacrolimus (MMF) treatment arm: MMF dose was initiated at 1 g b.i.d. (2 g/day). Adjustments were to be made for adverse events including, but not limited to, gastrointestinal intolerance and decrease in WBC. MMF trough or AUC was not used to adjust dosing. In this group, tacrolimus was initiated according to local practice. Tacrolimus dose was adjusted from Day 3 on to achieve a target whole blood trough concentration of 8 ng/mL to 12 ng/mL. From Month 2 until Month 6, target tacrolimus trough level was reduced to 7 - 10 ng/mL. After Month 6, target level of tacrolimus was reduced to 5 - 8 ng/mL.
  Interventions: Drug: mycophenolate mofetil and tacrolimus

INTERVENTIONS:
Drug: Everolimus and tacrolimus — Everolimus:
  * Dosage form: 0.75 mg, 0.25 mg, and 0.5 mg tablets
  * Dose: 1.5 mg per day
  * Frequency: 0.75 mg twice daily
  Tacrolimus:
  * Dose adjusted to maintain specific blood levels
  Arms: Everolimus (EVR) & low dose of tacrolimus
Drug: mycophenolate mofetil and tacrolimus — Mycophenolate mofetil: - Dose form: 250 mg capsule - Dose: 2g per day - Frequency: 1g twice daily Tacrolimus: - Dose adjusted to maintain specific blood levels
  Other Names: Active Comparator Control)
  Arms: Mycophenolate mofetil & standard dose tacrolimus

SUMMARY:
The purpose of this phase 3b study is to compare the safety and efficacy of everolimus with low dose tacrolimus to mycophenolate mofetil with standard dose tacrolimus in kidney transplant recipients.

ELIGIBILITY:
Inclusion criteria:

* Male or female renal recipients 18-70 years of age undergoing kidney transplantation, either primary or re-transplant;
* Recipient of a cadaveric, deceased donor (including expanded criteria donor organs and deceased donor organs after cardiac death), living unrelated or non-HLA identical living related donor kidney;
* Graft must be functional (producing greater than or equal to 100 ml of urine within 24 hours after transplantation) at time of randomization.

Exclusion criteria:

* Donor organ with a cold ischemic time > 30 hours;
* Males or females who produce less than 100 ml of urine in the first 24 hours post-transplantation;
* Males or females who are recipients of ABO incompatible transplants, or T cell, or B cell crossmatch positive transplant;
* Males or females with severe total hypercholesterolemia or total hypertriglyceridemia (Patients on lipid lowering treatment with controlled hyperlipidemia are acceptable);
* Males or females who have any surgical or any medical condition, such as severe diarrhea, active peptic ulcer disease, or uncontrolled diabetes mellitus, which in the opinion of the investigator, might alter the absorption, distribution, metabolism and/or excretion of study medication.

Other protocol related inclusion/exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 613 (Actual)
Dates: Start 2010-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (43):
- United States (42):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Orange, California
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Aurora, Colorado
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Worcester, Massachusetts
  - Novartis Investigative Site, Ann Arbor, Michigan
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, Royal Oak, Michigan
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Livingston, New Jersey
  - Novartis Investigative Site, Buffalo, New York
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Durham, North Carolina
  - Novartis Investigative Site, Greenville, North Carolina
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Harrisburg, Pennsylvania
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Fort Worth, Texas
  - Novartis Investigative Site, Galveston, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Lubbock, Texas
  - Novartis Investigative Site, Salt Lake City, Utah
  - Novartis Investigative Site, Burlington, Vermont
  - Novartis Investigative Site, Charlottesville, Virginia
  - Novartis Investigative Site, Norfolk, Virginia
  - Novartis Investigative Site, Richmond, Virginia
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Spokane, Washington
- Novartis Investigative Site, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Shihab F, Qazi Y, Mulgaonkar S, McCague K, Patel D, Peddi VR, Shaffer D. Association of Clinical Events With Everolimus Exposure in Kidney Transplant Patients Receiving Low Doses of Tacrolimus. Am J Transplant. 2017 Sep;17(9):2363-2371. doi: 10.1111/ajt.14215. Epub 2017 Mar 4. PMID 28141897

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total 738 participants were screened, and 613 were transplanted and randomized to treatment (n=309 to EVR+Low TAC dose and n=304 to MMF+Std TAC).
  EVR=Everolimus and low dose tacrolimus, and MMF=Mycophenolate mofetil and standard dose tacrolimus.
Groups:
- Everolimus and Low Dose Tacrolimus: Everolimus treatment arm: Therapeutic drug monitoring of everolimus and tacrolimus was mandatory throughout the study. From Day 5 onwards, the everolimus 0.75 mg b.i.d. dose was increased if the trough level was < 3 ng/mL, or reduced if the trough level was > 8 ng/mL. Tacrolimus was initiated according to local practice. In this treatment arm, the tacrolimus dose was adjusted from Day 3 onwards, to a target whole blood trough concentration of 4 ng/mL to 7 ng/mL. From Month 2 until Month 6, the target tacrolimus trough level was 3 ng/mL to 6 ng/mL. After Month 6, the tacrolimus dose was adjusted in order to achieve a target trough level of 2 ng/mL to 5 ng/mL.
- Mycophenolate Mofetil and Standard Dose Tacrolimus: MMF treatment arm: The MMF dose was initiated at 1 g b.i.d. (2 g/day). Adjustments were to be made for adverse events including, but not limited to, gastrointestinal intolerance and a decrease in WBC. MMF trough or AUC was not used to adjust dosing. In this group, tacrolimus was initiated according to local practice. The tacrolimus dose was adjusted from Day 3 on to achieve a target whole blood trough concentration of 8 ng/mL to 12 ng/mL. From Month 2 until Month 6, the target tacrolimus trough level was reduced to 7 - 10 ng/mL. After Month 6, the target level of tacrolimus was reduced to 5 - 8 ng/mL.
Period: Completed Study Medication
Arm/Group | Everolimus and Low Dose Tacrolimus | Mycophenolate Mofetil and Standard Dose Tacrolimus
Started | 309 | 304
Completed | 204 | 232
Not Completed | 105 | 72
Not completed — Adverse Event | 66 | 39
Not completed — Protocol Deviation | 9 | 8
Not completed — Withdrawal by Subject | 8 | 9
Not completed — Administrative problems | 7 | 5
Not completed — Unsatisfactory therapeutic effect | 7 | 0
Not completed — Abnormal test procedure | 4 | 0
Not completed — Graft loss | 2 | 5
Not completed — Death | 2 | 2
Not completed — Abnormal lab values | 0 | 2
Not completed — Subject no longer required study drug | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: Completed Study
Arm/Group | Everolimus and Low Dose Tacrolimus | Mycophenolate Mofetil and Standard Dose Tacrolimus
Started | 309 | 304
Completed | 293 (Completed study phase) | 282 (Completed study phase)
Not Completed | 16 | 22
Not completed — Withdrawal by Subject | 8 | 16
Not completed — Death | 6 | 5
Not completed — Missing | 2 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) consisted of all participants randomized after transplantation.
  *The discrepancy with the Ns is that there are 613 participants overall and 610 in the safety population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Everolimus and Low Dose Tacrolimus | Mycophenolate Mofetil and Standard Dose Tacrolimus | Total
Number analyzed (Participants) | 306 | 304 | 610
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.00 (13.34) | 48.4 (12.91) | 49.2 (13.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 102 | 203
  Male | 205 | 202 | 407
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 4
  Asian | 17 | 11 | 28
  Native Hawaiian or Other Pacific Islander | 3 | 1 | 4
  Black or African American | 70 | 74 | 144
  Caucasian | 196 | 201 | 397
  Other | 17 | 16 | 33
BMI [Mean (Standard Deviation); unit: kg/m˄2] — Body Mass Index
  kg/m˄2 | 27.7 (5.55) | 28.3 (5.13) | 28.0 (5.35)
Diabetic status at randomization [Number; unit: Participants] — 62 Insulin dependent + 49 Non-insulin dependent = 111 participants who were diabetic at randomization.
  Participants
    Yes | 111 | 95 | 206
    No | 195 | 209 | 404

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Incidence of Composite Efficacy Failure
Description: Efficacy failure rate used the composite endpoint of: (1) treated biopsy-proven acute rejection (BPAR)*, (2) graft loss**, (3) participant death or(4) loss to follow-up. *A treated BPAR was defined as a biopsy graded IA, IB, IIA, IIB, or III and which was treated with anti-rejection therapy. **Graft loss is defined as when the allograft was presumed lost on the day the participant started dialysis and was not able to subsequently be removed from dialysis.
Time Frame: 12 Months
Population: Full Analysis Set (FAS) consisted of all participants randomized after transplantation
Measure: Number; unit: Participants
Units Other Than Participants: Participants
Arm/Group | Everolimus and Low Dose Tacrolimus | Mycophenolate Mofetil and Standard Dose Tacrolimus
Number analyzed (Participants) | 309 | 304
Participants
  Composite Endpoint | 76 | 62
  Treated Biopsy-proven Acute rejection (BPAR) | 59 | 34
  Graft Loss | 4 | 12
  Death | 6 | 5
  Loss to follow up | 9 | 17

2. Secondary Outcome: Estimated Glomerular Filtration Rate (eGFR)
Description: Renal function was assessed by estimated Glomerular Filtration Rate (eGFR) using the Modification of Diet in Renal Disease (MDRD) formula. MDRD formula: GFR [mL/min/1.73m˄2] = 186.3*(C˄-1.154)*(A˄-0.203)*G*R. DEFINITIONS: C = serum concentration of creatinine [mg/dL]; A = age [years]; G = 0.742 when gender is female, otherwise G = 1; R = 1.21 when race is black, otherwise R = 1
Time Frame: 12 Months
Population: Full Analysis Set (FAS) consisted of all patients randomized after transplantation
Measure: Mean (Standard Deviation); unit: mL/min/1.73m˄2
Arm/Group | Everolimus and Low Dose Tacrolimus | Mycophenolate Mofetil and Standard Dose Tacrolimus
Number analyzed (Participants) | 309 | 304
mL/min/1.73m˄2 | 63.14 (22.042) | 63.06 (19.512)

3. Secondary Outcome: Number of Participants With Incidence of CMV (Viremia, Syndrome and Disease)
Description: Participants with incidence of CMV (viremia, syndrome and disease). CMV is cytomegalovirus.
Time Frame: 12 Months
Population: Safety Set (SS) consisted of all randomized participants who received at least 1 dose of study drug and had at least 1 post-baseline safety assessment. The statement that a patient had no adverse events constitutes a safety assessment. Those who received at least 1 dose of drug but had no post-treatment safety data of any kind are excluded from SS.
Measure: Number; unit: Participants
Units Other Than Participants: Participants
Arm/Group | Everolimus and Low Dose Tacrolimus | Mycophenolate Mofetil and Standard Dose Tacrolimus
Number analyzed (Participants) | 306 | 304
Participants
  CMV syndrome event | 9 | 13
  Lab evidence of CMV Viremia | 7 | 10
  CMV Disease | 2 | 8

4. Secondary Outcome: Number of Participants With Incidence Rates of BKV Viremia, BKV Viruria, or BKV Nephropathy
Description: Participants with Incidence of BKV (viremia, viruria, or nephropathy). BKV is Polyomavirus type BK.
Time Frame: 12 Months
Population: as for outcome 3
Measure: Number; unit: Participants
Units Other Than Participants: Participants
Arm/Group | Everolimus and Low Dose Tacrolimus | Mycophenolate Mofetil and Standard Dose Tacrolimus
Number analyzed (Participants) | 306 | 304
Participants
  Lab evidence of BKV Viremia | 19 | 27
  Lab evidence of BKV Viruria | 19 | 15
  BKV Disease (Nephropathy) | 5 | 5

5. Secondary Outcome: Number of Participants With Incidence of New Onset of Diabetes Mellitus
Description: Incidence of new onset diabetes mellitus defined as non-diabetic patients before transplantation, who are receiving glucose lowering treatment for more than 30 days post-transplant, or with a random plasma glucose ≥200 mg dL (11.1 mmol/L) with 2 fasting plasma glucose values ≥126 mg/dL (7 mmol/L)
Time Frame: 12 Months
Population: as for outcome 3
Measure: Number; unit: Participants
Units Other Than Participants: Participants
Arm/Group | Everolimus and Low Dose Tacrolimus | Mycophenolate Mofetil and Standard Dose Tacrolimus
Number analyzed (Participants) | 306 | 304
Participants
  Any New Onset Diabetes | 25 | 22
  randomGlucose≥200mg/dL w/2 fastingGlucose≥126mg/dL | 15 | 12
  Concomitant Diabetes medicine for 30 days or more | 13 | 14

6. Secondary Outcome: Number of Participants With Incidence of Proteinuria Events
Description: Number of participants with Incidence of proteinuria events indicating chronic kidney disease
Time Frame: Baseline and 12 Months
Population: as for outcome 3
Measure: Number; unit: Participants
Units Other Than Participants: Participants
Arm/Group | Everolimus and Low Dose Tacrolimus | Mycophenolate Mofetil and Standard Dose Tacrolimus
Number analyzed (Participants) | 306 | 304
Participants
  Baseline: Proteinuria (>=300 mg/g) | 243 | 250
  Month 12, Day 316-450: Proteinuria (>=300 mg/g) | 36 | 35

7. Secondary Outcome: Number of Participants With Incidence of Adverse Events, Serious Adverse Events, and Tacrolimus-associated Adverse Events
Description: Incidence of adverse events, serious adverse events, and tacrolimus-associated adverse events by System Organ Class
Time Frame: 12 Months
Population: as for outcome 3
Measure: Number; unit: Participants
Units Other Than Participants: Participants
Arm/Group | Everolimus and Low Dose Tacrolimus | Mycophenolate Mofetil and Standard Dose Tacrolimus
Number analyzed (Participants) | 306 | 304
Participants
  Any system organ class | 303 | 302
  Metabolism and nutrition disorders | 266 | 263
  Gastrointestinal disorders | 233 | 247
  Injury, poisoning and procedural complications | 223 | 202
  General disorders &administration site conditions | 199 | 177
  Infections and infestations | 184 | 196
  Investigations | 150 | 143
  Renal and urinary disorders | 141 | 160
  Vascular disorders | 131 | 121
  Blood and lymphatic system disorders | 130 | 163
  Nervous system disorders | 125 | 150
  Respiratory, thoracic and mediastinal disorders | 122 | 134
  Musculoskeletal and connective tissue disorders | 110 | 114
  Skin and subcutaneous tissue disorders | 109 | 108
  Psychiatric disorders | 96 | 106
  Reproductive system and breast disorders | 56 | 40
  Cardiac disorders | 51 | 47
  Eye disorders | 26 | 36
  Immune system disorders | 13 | 11
  Endocrine disorders | 12 | 8
  Neoplasms benign,malignant,other incl cysts/polyps | 10 | 15
  Ear and labyrinth disorders | 7 | 11
  Hepatobiliary disorders | 6 | 3
  Surgical and medical procedures | 2 | 0
  Congenital, familial and genetic disorders | 0 | 6
  Social circumstances | 0 | 1

ADVERSE EVENTS:
Groups:
- Everolimus and Low Dose Tacrolimus: Therapeutic drug monitoring of everolimus and tacrolimus was mandatory throughout the study. From Day 5 onwards, the everolimus 0.75 mg b.i.d. dose was increased if the trough level was < 3 ng/mL, or reduced if the trough level was > 8 ng/mL. Tacrolimus was initiated according to local practice. In this treatment arm, the tacrolimus dose was adjusted from Day 3 onwards, to a target whole blood trough concentration of 4 ng/mL to 7 ng/mL. From Month 2 until Month 6, the target tacrolimus trough level was 3 ng/mL to 6 ng/mL. After Month 6, the tacrolimus dose was adjusted in order to achieve a target trough level of 2 ng/mL to 5 ng/mL.
- Mycophenolate Mofetil and Standard Dose Tacrolimus: The MMF dose was initiated at 1 g b.i.d. (2 g/day). Adjustments were to be made for adverse events including, but not limited to, gastrointestinal intolerance and a decrease in WBC. MMF trough or AUC was not used to adjust dosing. In this group, tacrolimus was initiated according to local practice. The tacrolimus dose was adjusted from Day 3 on to achieve a target whole blood trough concentration of 8 ng/mL to 12 ng/mL. From Month 2 until Month 6, the target tacrolimus trough level was reduced to 7 - 10 ng/mL. After Month 6, the target level of tacrolimus was reduced to 5 - 8 ng/mL.
Arm/Group | Everolimus and Low Dose Tacrolimus | Mycophenolate Mofetil and Standard Dose Tacrolimus
Serious Adverse Events (participants affected / at risk) | 154/306 | 142/304
Other Adverse Events (participants affected / at risk) | 302/306 | 299/304
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus and Low Dose Tacrolimus (N=306) | Mycophenolate Mofetil and Standard Dose Tacrolimus (N=304)
Anaemia (Blood and lymphatic system disorders) | 3 | 4
Bandaemia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 2 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 3
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 4
Atrial fibrillation (Cardiac disorders) | 2 | 3
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 2
Cardiac failure congestive (Cardiac disorders) | 5 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 2
Sinus tachycardia (Cardiac disorders) | 1 | 0
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 | 1
Congenital renal cyst (Congenital, familial and genetic disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 2 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 1
Diabetic gastroparesis (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 8
Erosive oesophagitis (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 2
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 1
Internal hernia (Gastrointestinal disorders) | 1 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 7 | 4
Neutropenic colitis (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Oral pain (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Peptic ulcer (Gastrointestinal disorders) | 1 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 1
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0
Tongue ulceration (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 8 | 7
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 2 | 5
Chills (General disorders) | 1 | 1
Device malfunction (General disorders) | 1 | 1
Fatigue (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 0 | 1
Generalised oedema (General disorders) | 1 | 1
Hernia (General disorders) | 2 | 1
Impaired healing (General disorders) | 3 | 0
Irritability (General disorders) | 0 | 1
Medical device complication (General disorders) | 0 | 1
Oedema (General disorders) | 2 | 0
Oedema peripheral (General disorders) | 3 | 2
Pyrexia (General disorders) | 13 | 11
Rebound effect (General disorders) | 0 | 1
Sluggishness (General disorders) | 0 | 1
Kidney transplant rejection (Immune system disorders) | 1 | 1
Transplant rejection (Immune system disorders) | 1 | 1
Adenovirus infection (Infections and infestations) | 0 | 1
BK virus infection (Infections and infestations) | 1 | 1
Bacteraemia (Infections and infestations) | 1 | 4
Bacterial pyelonephritis (Infections and infestations) | 0 | 2
Bronchitis (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 6 | 3
Cellulitis of male external genital organ (Infections and infestations) | 0 | 1
Cerebral fungal infection (Infections and infestations) | 1 | 0
Clostridial infection (Infections and infestations) | 3 | 3
Clostridium difficile colitis (Infections and infestations) | 0 | 2
Cystitis (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 5
Cytomegalovirus viraemia (Infections and infestations) | 1 | 1
Device related infection (Infections and infestations) | 1 | 1
Enterococcal bacteraemia (Infections and infestations) | 1 | 0
Escherichia bacteraemia (Infections and infestations) | 1 | 1
Escherichia sepsis (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 2 | 0
Gangrene (Infections and infestations) | 2 | 2
Gastroenteritis (Infections and infestations) | 3 | 2
Gastroenteritis clostridial (Infections and infestations) | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 3 | 3
Incision site infection (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Lung infection pseudomonal (Infections and infestations) | 1 | 0
Mastitis (Infections and infestations) | 1 | 0
Meningitis cryptococcal (Infections and infestations) | 0 | 1
Metapneumovirus infection (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 13 | 7
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pneumonia cryptococcal (Infections and infestations) | 0 | 1
Pneumonia cytomegaloviral (Infections and infestations) | 0 | 1
Polyomavirus-associated nephropathy (Infections and infestations) | 0 | 2
Post procedural cellulitis (Infections and infestations) | 1 | 0
Pseudomonal bacteraemia (Infections and infestations) | 1 | 0
Pulmonary mycosis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 6 | 4
Sepsis (Infections and infestations) | 1 | 2
Septic shock (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 22 | 24
Urinary tract infection bacterial (Infections and infestations) | 1 | 2
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0
Urinary tract infection pseudomonal (Infections and infestations) | 0 | 1
Urinary tract infection staphylococcal (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 5 | 7
Viraemia (Infections and infestations) | 0 | 2
Viral infection (Infections and infestations) | 1 | 1
Wound infection (Infections and infestations) | 4 | 2
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 | 1
Complications of transplant surgery (Injury, poisoning and procedural complications) | 1 | 0
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 4 | 4
Device dislocation (Injury, poisoning and procedural complications) | 0 | 1
Graft complication (Injury, poisoning and procedural complications) | 2 | 1
Graft dysfunction (Injury, poisoning and procedural complications) | 9 | 8
Graft loss (Injury, poisoning and procedural complications) | 2 | 3
Graft thrombosis (Injury, poisoning and procedural complications) | 2 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Incision site complication (Injury, poisoning and procedural complications) | 1 | 0
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 2 | 1
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Medical device complication (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Perinephric collection (Injury, poisoning and procedural complications) | 3 | 1
Perirenal haematoma (Injury, poisoning and procedural complications) | 3 | 1
Post procedural discharge (Injury, poisoning and procedural complications) | 1 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 0 | 1
Post procedural urine leak (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1
Renal haematoma (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 2 | 2
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 2
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Urinary anastomotic leak (Injury, poisoning and procedural complications) | 1 | 0
Vascular graft complication (Injury, poisoning and procedural complications) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 3 | 1
Blood creatine increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 10 | 14
Blood glucose increased (Investigations) | 0 | 1
Electrocardiogram ST segment elevation (Investigations) | 1 | 0
Escherichia test positive (Investigations) | 1 | 0
Transaminases increased (Investigations) | 2 | 0
Urine output decreased (Investigations) | 1 | 2
White blood cell count increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 6 | 5
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 7
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 2
Fluid overload (Metabolism and nutrition disorders) | 6 | 1
Fluid retention (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 6
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 6
Hyperosmolar state (Metabolism and nutrition disorders) | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone giant cell tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pleural mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 1
Embolic stroke (Nervous system disorders) | 0 | 1
Encephalitis (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Unresponsive to stimuli (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 1
Disorientation (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 3 | 3
Psychotic disorder (Psychiatric disorders) | 0 | 1
Bladder spasm (Renal and urinary disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1
Focal segmental glomerulosclerosis (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 2 | 5
Hydronephrosis (Renal and urinary disorders) | 3 | 6
Hydroureter (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Obstructive uropathy (Renal and urinary disorders) | 2 | 0
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal aneurysm (Renal and urinary disorders) | 1 | 0
Renal artery stenosis (Renal and urinary disorders) | 2 | 2
Renal artery thrombosis (Renal and urinary disorders) | 1 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0
Renal cyst ruptured (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 2 | 1
Renal failure acute (Renal and urinary disorders) | 7 | 16
Renal failure chronic (Renal and urinary disorders) | 1 | 1
Renal impairment (Renal and urinary disorders) | 3 | 0
Renal injury (Renal and urinary disorders) | 1 | 1
Renal pain (Renal and urinary disorders) | 0 | 1
Renal tubular necrosis (Renal and urinary disorders) | 4 | 2
Renal vein thrombosis (Renal and urinary disorders) | 1 | 2
Ureteric stenosis (Renal and urinary disorders) | 2 | 3
Urethral stenosis (Renal and urinary disorders) | 1 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 4
Urinary retention (Renal and urinary disorders) | 0 | 3
Urinary tract obstruction (Renal and urinary disorders) | 1 | 1
Urinoma (Renal and urinary disorders) | 2 | 0
Vesicoureteric reflux (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Pelvic haematoma (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 7 | 0
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Pyelotomy (Surgical and medical procedures) | 1 | 0
Arteriovenous fistula (Vascular disorders) | 1 | 1
Blood pressure inadequately controlled (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 4 | 5
Extremity necrosis (Vascular disorders) | 0 | 1
Extrinsic iliac vein compression (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 1
Haemorrhage (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 7 | 3
Hypertensive crisis (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 0 | 3
Iliac artery thrombosis (Vascular disorders) | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 2 | 0
Lymphocele (Vascular disorders) | 7 | 4
Orthostatic hypotension (Vascular disorders) | 0 | 2
Peripheral vascular disorder (Vascular disorders) | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 2 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
Venous stenosis (Vascular disorders) | 0 | 2
Venous thrombosis limb (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus and Low Dose Tacrolimus (N=306) | Mycophenolate Mofetil and Standard Dose Tacrolimus (N=304)
Anaemia (Blood and lymphatic system disorders) | 83 | 67
Leukocytosis (Blood and lymphatic system disorders) | 22 | 31
Leukopenia (Blood and lymphatic system disorders) | 27 | 65
Neutropenia (Blood and lymphatic system disorders) | 7 | 24
Thrombocytopenia (Blood and lymphatic system disorders) | 22 | 16
Tachycardia (Cardiac disorders) | 22 | 20
Abdominal distension (Gastrointestinal disorders) | 17 | 22
Abdominal pain (Gastrointestinal disorders) | 29 | 35
Constipation (Gastrointestinal disorders) | 119 | 120
Diarrhoea (Gastrointestinal disorders) | 74 | 122
Dyspepsia (Gastrointestinal disorders) | 20 | 23
Flatulence (Gastrointestinal disorders) | 10 | 19
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 18 | 28
Nausea (Gastrointestinal disorders) | 111 | 134
Vomiting (Gastrointestinal disorders) | 45 | 64
Fatigue (General disorders) | 58 | 52
Oedema (General disorders) | 32 | 28
Oedema peripheral (General disorders) | 113 | 88
Pyrexia (General disorders) | 41 | 47
BK virus infection (Infections and infestations) | 32 | 41
Nasopharyngitis (Infections and infestations) | 13 | 20
Upper respiratory tract infection (Infections and infestations) | 28 | 33
Urinary tract infection (Infections and infestations) | 49 | 68
Graft dysfunction (Injury, poisoning and procedural complications) | 35 | 32
Incision site pain (Injury, poisoning and procedural complications) | 46 | 54
Procedural pain (Injury, poisoning and procedural complications) | 93 | 94
Blood creatinine increased (Investigations) | 49 | 41
Weight increased (Investigations) | 20 | 14
Decreased appetite (Metabolism and nutrition disorders) | 6 | 23
Dehydration (Metabolism and nutrition disorders) | 17 | 18
Diabetes mellitus (Metabolism and nutrition disorders) | 32 | 30
Fluid overload (Metabolism and nutrition disorders) | 21 | 23
Hypercalcaemia (Metabolism and nutrition disorders) | 12 | 17
Hyperglycaemia (Metabolism and nutrition disorders) | 75 | 81
Hyperkalaemia (Metabolism and nutrition disorders) | 93 | 81
Hyperlipidaemia (Metabolism and nutrition disorders) | 71 | 31
Hyperphosphataemia (Metabolism and nutrition disorders) | 23 | 25
Hypocalcaemia (Metabolism and nutrition disorders) | 46 | 40
Hypoglycaemia (Metabolism and nutrition disorders) | 20 | 23
Hypokalaemia (Metabolism and nutrition disorders) | 56 | 54
Hypomagnesaemia (Metabolism and nutrition disorders) | 102 | 124
Hyponatraemia (Metabolism and nutrition disorders) | 11 | 21
Hypophosphataemia (Metabolism and nutrition disorders) | 108 | 94
Metabolic acidosis (Metabolism and nutrition disorders) | 35 | 39
Vitamin D deficiency (Metabolism and nutrition disorders) | 21 | 25
Arthralgia (Musculoskeletal and connective tissue disorders) | 31 | 23
Back pain (Musculoskeletal and connective tissue disorders) | 21 | 23
Muscle spasms (Musculoskeletal and connective tissue disorders) | 15 | 20
Pain in extremity (Musculoskeletal and connective tissue disorders) | 28 | 24
Dizziness (Nervous system disorders) | 26 | 36
Headache (Nervous system disorders) | 44 | 53
Hypoaesthesia (Nervous system disorders) | 17 | 9
Tremor (Nervous system disorders) | 51 | 86
Anxiety (Psychiatric disorders) | 17 | 33
Insomnia (Psychiatric disorders) | 68 | 71
Dysuria (Renal and urinary disorders) | 24 | 25
Haematuria (Renal and urinary disorders) | 30 | 33
Proteinuria (Renal and urinary disorders) | 31 | 19
Renal tubular necrosis (Renal and urinary disorders) | 20 | 19
Urinary retention (Renal and urinary disorders) | 17 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 28 | 43
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 40 | 49
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 23 | 24
Acne (Skin and subcutaneous tissue disorders) | 20 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 18
Pruritus (Skin and subcutaneous tissue disorders) | 32 | 32
Rash (Skin and subcutaneous tissue disorders) | 24 | 12
Hypertension (Vascular disorders) | 64 | 71
Hypotension (Vascular disorders) | 25 | 29

LIMITATIONS AND CAVEATS:
HLA mismatches ≥3, everolimus group 261 vs MMF group 240

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial; or disclosure of the trial results in their entirety.